CLINICAL TRIAL: NCT03753217
Title: Assessment of the Depth of Anesthesia During Intravenous Anesthesia: Comparison of the Bispectral Index Monitor and the qCON Monitor.
Brief Title: Comparison of Two Electroencephalograms (EEG) Monitors in Patients Undergoing General Intravenous Anesthesia
Acronym: Bis-qCON-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016/57
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-08

CONDITIONS: General Anesthesia
Keywords: Anesthesia Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- qCON Monitor (Experimental): Simultaneous measurement of BIS and qCON
  Interventions: Device: qCON Monitor

INTERVENTIONS:
Device: qCON Monitor — supervision by qCON monitor of the depth of anesthesia

SUMMARY:
Quantium Medical Company has an ElectroEncephalograph-based (EEG-based) algorithm with two outputs: qCON for unconsciousness and qNOX for anti-nociception. qCON, is designed to provide information about the depth of the hypnotic state, similar to that provided by the BIS™.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years,
* Patients affiliated to a national insurance scheme or benefiting from such a program,
* Patients having given their written consent,
* Patients that must benefit from a general anesthesia by intravenous drugs (propofol and remifentanil),
* For the patients taken care in ambulatory surgery, having a telephone and agreeing to communicate their phone number.

Exclusion Criteria:

* Pregnant or breast-feeding Women,
* Patients having a limit of use of the Bispectral Index (BIS) or qCON monitors,
* Patients having a contraindication to Propofol and/or to Remifentanil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
qCON monitoring during maintenance of anesthesia | Up to 10 hours
  Measurement of qCON values during maintenance of anesthesia
BIS monitoring during maintenance of anesthesia | Up to 10 hours
  Measurement of BIS values during maintenance of anesthesia

SECONDARY OUTCOMES:
qCON monitoring during induction of anesthesia | One day
  Measurement of qCON values during induction of anesthesia
BIS monitoring during induction of anesthesia | One day
  Measurement of BIS values during induction of anesthesia
qCON monitoring during recovery of anesthesia | One day
  Measurement of qCON values during recovery of anesthesia
BIS monitoring during recovery of anesthesia | One day
  Measurement of BIS values during recovery of anesthesia
Burst Suppression ratio retrieved by qCON monitoring | One day
  Measurement of Burst Suppression ratio values during anesthesia
Burst Suppression ratio retrieved by BIS monitoring | One day
  Measurement of Burst Suppression ratio values during anesthesia
qNOX monitoring during anesthesia | One day
  Measurement of qNOX values during anesthesia
Periods of loss of signal of qCON | One day
  Measurement of qCON values during anesthesia
Periods of loss of signal of BIS | One day
  Measurement of BIS values during anesthesia
Intraoperative memorising | One day
  Questionnaire for assessment of memorising of surgery by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD PhD, Study Director — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No